CLINICAL TRIAL: NCT04335487
Title: Internet-Delivered Cognitive Behaviour Therapy for PTSD Among Public Safety Personnel: Open Cohort Preference Trial for Transdiagnostic or Disorder-Specific Therapy
Brief Title: Internet-Delivered Cognitive Behaviour Therapy for PTSD Among Public Safety Personnel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Government of Canada (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-157b
Record Dates: First submitted 2020-03-31; First posted 2020-04-06 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Posttraumatic Stress; Depression; Anxiety
Keywords: Internet; Cognitive Behavioral Therapy; Telemedicine
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Preference trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICBT for PTSD Tailored for PSP (Experimental): Therapist-guided, Internet-delivered cognitive behavioral therapy for PTSD tailored specifically for Canadian public safety personnel.
  Interventions: Behavioral: PSP PTSD Course
- Transdiagnostic ICBT Tailored for PSP (Experimental): Therapist-guided, transdiagnostic Internet-delivered cognitive behavioral therapy tailored specifically for Canadian public safety personnel.
  Interventions: Behavioral: PSP Wellbeing Course

INTERVENTIONS:
Behavioral: PSP PTSD Course — A tailored ICBT intervention designed to treat symptoms of PTSD will be delivered to public safety personnel. Clients will be offered once a week support, but support can be increased to twice a week support if PSP request extra support. The intervention is designed to be completed in 8 weeks, but clients will be able to extend their treatment by an additional 8 weeks (i.e., up to 16 weeks in total).
  Arms: ICBT for PTSD Tailored for PSP
Behavioral: PSP Wellbeing Course — A tailored ICBT intervention designed to treat symptoms of depression, anxiety, or PTSD will be delivered to public safety personnel. Clients will be offered once a week support, but support can be increased to twice a week support if PSP request extra support. The intervention is designed to be completed in 8 weeks, but clients will be able to extend their treatment by an additional 8 weeks (i.e., up to 16 weeks in total).
  Arms: Transdiagnostic ICBT Tailored for PSP

SUMMARY:
This study evaluates two Internet-delivered cognitive behavioural therapy (ICBT) interventions: one for symptoms of posttraumatic stress disorder (PTSD) and one for symptoms of anxiety, depression, and PTSD. Both interventions have been tailored for Canadian public safety personnel (PSP). Outcomes of interest include preference for disorder-specific or transdiagnostic care, engagement with the interventions, changes in symptoms and functioning, and strengths and limitations of implementing ICBT with Canadian PSP.

DETAILED DESCRIPTION:
Background:

Public Safety Personnel (PSP) is a term that broadly encompasses personnel who ensure the safety and security of Canadians across jurisdictions, including, but not necessarily limited to, border services personnel, correctional employees, firefighters (career and volunteer), operational and intelligence personnel, paramedics, police officers, public safety communications officials (e.g., call centre operators/dispatchers), and search and rescue personnel. As a function of their vocations, PSP are frequently exposed to potentially psychologically traumatic events (e.g., threatened or actual physical assaults, sexual violence, fires, and explosions) and are at risk of posttraumatic stress injuries. Results from a recent survey with a large Canadian PSP sample showed 44.5% screened positive for one or more mental health disorders, which is much higher than the 10.1% diagnostic rate among the Canadian general public. The study showed that 23.2% of Canadian PSP screened positive for PTSD, and 25.7% screened positive for two or more mental disorders. For many Canadian PSP, access to in-person evidence-based care is impeded for several logistical reasons, including distance from services, long waiting lists, difficulty navigating services, and the cost of treatment. PSP also face attitudinal barriers, including concerns about stigma, discomfort admitting to needing help, distrust of service providers, and lack of awareness of their need for help.

Internet-delivered cognitive behaviour therapy (ICBT) represents a convenient method for PSP to access care for mental health concerns, such as posttraumatic stress. In ICBT, clients receive access to standardized lessons that provide the same information and skills as traditional face-to-face CBT. In addition to weekly lessons, clients are encouraged to complete homework assignments to facilitate learning. Research shows that ICBT is effective at reducing symptoms of posttraumatic stress, and there is also evidence that the findings of research trials translate into routine clinic settings.

Research Purpose:

The current research project is designed to compare preference for disorder-specific program for PTSD (PSP PTSD Course) versus a transdiagnostic program for depression, anxiety, and PTSD (PSP Wellbeing Course); both courses have been adapted to be specific to PSP (e.g., case examples are relevant to PSP). The study will also examine engagement and outcomes of the courses. The current study outcome variables will include: 1) usage of both courses among Canadian PSP who are informed about the courses (e.g., # enrolling, completion rates); 2) symptoms of depression, anxiety, and PTSD, as well as secondary outcome measures (e.g., treatment satisfaction, disability) from PSP participants measured at 8, and 26 week follow-up; and 3) strengths and challenges of both courses when offered to PSP. In order to take part, PSP will first complete an online questionnaire and telephone screening to assess whether they meet the following inclusion criteria: 1) 18 years of age or older; 2) resident of the Canadian provinces of Saskatchewan, Quebec, Nova Scotia, New Brunswick, Prince Edward Island, or Ontario; 3) endorsing symptoms of posttraumatic stress, but not high suicide risk or recent suicide attempts in the past year; 4) able to access and comfortable using computers and the internet; 5) not seeking help primarily for alcohol and or drugs, bipolar disorder, or psychotic symptoms; and 6) willing to provide an emergency contact unless the participant does not have a physician and the clinician assesses the need for an emergency contact as low during the telephone screening. Eligible participants will be invited to choose either of the two courses. Both courses will be delivered by trained providers with graduate training in psychology or social work or graduate students under supervision. The programs were first offered in Saskatchewan and later translated into French and offered to PSP in Quebec, Nova Scotia, New Brunswick, Prince Edward Island, and Ontario. The primary research questions to be answered include:

1. ENGAGEMENT: How many PSP will enroll in and complete each course? Of note, we had initially planned to investigate how often PSP engage with therapists and how often PSP extend support beyond 8 weeks, but unforeseen system-related challenges rendered these research questions difficult to investigate in an unintrusive manner, so we have abandoned these research questions.
2. OUTCOMES: What will be the impact of the each course on symptom improvement and functioning at 8, 26, and 52 weeks post-enrollment? What factors will predict outcomes (e.g., symptom severity, demographics, engagement)? Please note: Effective December 2024, we have discontinued data collection at the 52-week post-enrollment mark. This decision was made due to low response rates at this time point and limited resources available to enhance enrollment efforts.
3. IMPLEMENTATION: What are stakeholder experiences, positive and negative, with each course? What are the suggested improvements to ICBT to meet the needs of PSP?

Significance:

This project will provide information that will inform future use of ICBT to assist PSP with symptoms of depression, anxiety, and PTSD.

Deviations from Original Trial Protocol:

We have made several changes to our methods since releasing our original trial protocol: (a) expanding access to this study to PSP residing in the Canadian provinces of Saskatchewan, Quebec, Nova Scotia, New Brunswick, Prince Edward Island, and Ontario due to interest from these provinces; (b) replacing the Sheehan Disability Scale with the Work and Social Adjustment Scale because we were unable to obtain permission to use the former; (c) removing a clinical interview from our planned outcome measures (Section H of the Mini International Neuropsychiatric Interview) due to lack of resources; (d) removing two questionnaires assessing exposure to potentially psychologically traumatic events (the Life Events Checklist for DSM-5 and a bespoke questionnaire inquiring about the worst event ever experienced) to reduce the burden of questionnaires on clients; (e) limiting our administration of outcome measures between 9 and 16 weeks post-enrollment to clients who are still engaged in treatment at those timepoints (i.e., rather than to all clients at those timepoints) to reduce the burden of questionnaires on clients; (f) extending the trial and increasing our estimated enrollment from 50 participants to 300 participants to better address our research objectives and because we have been able to expand recruitment efforts across several provinces; (g) replacing the 6-item version of the Social Interaction Anxiety Scale and the 6-item version of the Social Phobia Scale (SIAS-6/SPS-6) with the Mini Social Phobia Inventory (Mini-SPIN); (h) replacing the Panic Disorder Severity Scale-Self Report (PDSS-SR) with a 2-item version of the same measure; (i) replacing the Drug Use Disorders Identification Test (DUDIT) with the condensed version (DUDIT-C); (j) adding the abbreviated clinical version of the Moral Injury Outcome Scale (MIOS-AC); and (k) no longer administering measures at week 52."

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* residing in Saskatchewan for the duration of the intervention
* endorsing symptoms of post-traumatic stress
* able to access a computer and internet service
* willing to provide a physician as emergency contact

Exclusion Criteria:

* high suicide risk
* suicide attempt or hospitalization in the last year
* primary problems with psychosis, alcohol or drug problems, or mania
* currently receiving regular psychological treatment
* concerns about ICBT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in posttraumatic stress | screening and 8, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  PTSD Checklist for DSM-5 (PCL-5). Higher total scores indicate greater severity of posttraumatic stress. Scores range from 0 to 80. This measure is administered at screening and 8, 26, and 52 weeks.
  Abbreviated PTSD Checklist - Civilian Version (PCL-C). Six items. Higher total scores indicate greater severity of posttraumatic stress. Scores range from 5 to 30. This measure is administered to help clinicians track progress and is administered weekly at weeks 1 to 7 and 9 to 16 post-enrollment if clients are still engaged in treatment at those timepoints.

SECONDARY OUTCOMES:
Change in depression | screening and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Patient Health Questionnaire - 9 Item (PHQ-9). Higher total scores indicate greater severity of depression. Scores range from 0 to 27. Note: this measure is only administered at 9 through 16 weeks for clients who are still engaged in treatment at those timepoints.
Change in anxiety | screening and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Generalized Anxiety Disorder - 7 Item (GAD-7). Higher total scores indicate greater severity of anxiety. Scores range from 0 to 21. Note: this measure is only administered at 9 through 16 weeks for clients who are still engaged in treatment at those timepoints.
Change in panic symptoms | screening and 8, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Panic Disorder Severity Scale-Self Report, (PDSS-SR), 2-item version. Higher total scores indicate greater severity of panic symptoms. Scores range from 0 to 8. Note: this measure replaced the full PDSS-SR on October 6th, 2023.
Change in social anxiety | screening and 8, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Mini Social Phobia Inventory (Mini-SPIN). Higher total scores indicate greater severity of social anxiety. Scores range from 0 to 12. Note: this measure was added on October 6th, 2023.
Change in anger | screening and 8, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Dimensions of Anger Reactions (DAR-5) scale. Higher total scores indicate greater severity of anger problems. Scores range from 0 to 20.
Alcohol use | screening
  Alcohol Use Disorders Identification Test (AUDIT). Higher scores indicate greater alcohol consumption and alcohol-related problems. Scores ranger from 0 to 40.
Drug use | screening
  Drug Use Disorders Identification Test-C (DUDIT-C). Higher scores indicate greater drug use and drug-related problems. Scores ranger from 0 to 16. Note: this measure replaced the full DUDIT in December 2024.
Change in functioning | screening and 4, 8, 12, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Work and Social Adjustment Scale (WSAS). Higher total scores indicate a greater degree of impairment. Total scores range from 0 to 40. Note: this measure is only administered at 12 weeks for clients who are still engaged in treatment at this timepoint. Note: this measure replaced the Sheehan Disability Scale (SDS).
Change in use of health services | screening and 8, 26, and 52 weeks
  Health Service Use Questionnaire is a bespoke questionnaire that assesses the use of health services for mental health problems.
Treatment satisfaction | week 8
  Treatment Satisfaction Questionnaire. A bespoke questionnaire consisting of 32 items with varying response formats measuring treatment satisfaction and perceived treatment credibility. Items are not designed to be combined into a unitary measure.
Working alliance | week 8
  Working Alliance Inventory - Short Revised (WAI-SR). Higher scores indicate greater working alliance. Scores in three distinct domains of working alliance each range from 4 to 20.
Engagement and homework compliance | 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 weeks.
  Homework Reflection. A bespoke questionnaire consisting of 8 items with varying response formats, designed to measure engagement with treatment tasks and help alert therapists to any challenges clients face. Items are not designed to be combined into a unitary measure. Note: this measure is only administered at 9, 10, 11, and 12 weeks for clients who are still engaged in treatment at those timepoints.
Change in Moral Injury | screening, 8 and 26 weeks.
  Moral Injury Outcome Scale - Abbreviated Winter Campaign version. High total scores indicate greater levels of current moral injury. Scores range from 0 - 56. Note: this measure was added in December 2024

CONTACTS AND LOCATIONS:
Overall Officials: Heather D Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Department of Psychology and Collaborative Centre for Justice and Safety, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Price JA, McCall HC, Demyen SA, Spencer SM, Katz BM, Clairmont AP, Hadjistavropoulos HD. Optimization of Internet-Delivered Cognitive Behavioral Therapy for Canadian Leaders Within Public Safety: Qualitative Study. J Med Internet Res. 2025 Apr 17;27:e72321. doi: 10.2196/72321. PMID 40245389
- See also: Additional information about PSPNET. — https://www.pspnet.ca/